CLINICAL TRIAL: NCT01486589
Title: Risk Stratification in the Emergency Room by Cardiac Autonomic Function
Brief Title: Cardiac Autonomic Function For Risk Stratification in the Emergency Room
Acronym: PREDICT-ER
Status: Completed | Type: Observational
Sponsor: Thebiosignals.com (Other)
Responsible Party: Principal Investigator, Axel Bauer, Prof. Dr. Axel Bauer, University Hospital Tuebingen
Other Study IDs: 577/2011BO1
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Autonomic Nervous System Activity
Keywords: emergency care; cardiac autonomic function; deceleration capacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to test the hypothesis that impaired cardiac autonomic function predicts adverse outcome in unselected patients presenting in the emergency ward.

ELIGIBILITY:
Inclusion Criteria:

- presenting at the emergency department of the University Hospital of Tübingen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients presenting at the emergency department of the University Hospital of Tübingen
Sampling Method: Non-Probability Sample
Enrollment: 6521 (Actual)
Dates: Start 2010-10; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | 10 days

SECONDARY OUTCOMES:
Cardiac mortality | 10 days
transfer to intensive care unit | 10 days
hospital discharge | 48 hours
duration of hospital stay | within 30 days
costs of health care | 30 days
180 day mortality | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Universitätsklinik Tübingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Eick C, Duckheim M, Groga-Bada P, Klumpp N, Mannes S, Zuern CS, Gawaz M, Rizas KD, Bauer A. Point-of-care testing of cardiac autonomic function for risk assessment in patients with suspected acute coronary syndromes. Clin Res Cardiol. 2017 Sep;106(9):686-694. doi: 10.1007/s00392-017-1104-3. Epub 2017 Mar 22. PMID 28331988
- [Derived] Eick C, Rizas KD, Meyer-Zurn CS, Groga-Bada P, Hamm W, Kreth F, Overkamp D, Weyrich P, Gawaz M, Bauer A. Autonomic nervous system activity as risk predictor in the medical emergency department: a prospective cohort study. Crit Care Med. 2015 May;43(5):1079-86. doi: 10.1097/CCM.0000000000000922. PMID 25738854